CLINICAL TRIAL: NCT02866487
Title: Lung Fluid and Peripheral Blood Neutrophil IL-5 Surface Receptor in Children With Asthma
Acronym: NAIL-5
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Willliam Gerald Teague, Ivy Foundation Distinguished Professor of Pediatrics, University of Virginia
Other Study IDs: NAIL-5
Record Dates: First submitted 2016-07-28; First posted 2016-08-15 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood, bronchoalveolar (BAL) fluid, nasal wash/absorbent pad fluid, and nasal scraping epithelial cells will be collected for study analyses with leftover samples banked for future research
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthmatics: 0-5 years of age: Intermittent cough, wheeze, chest symptoms AND one or more of the following: Eczema Eosinophilia Elevated total IgE Positive family history
  6-17 years of age: Physician diagnosis Current treatment with one or more asthma medications Recurrent episodes of cough, wheeze, chest discomfort, pain
  Interventions: Procedure: Bronchoscopy
- Age-Similar Non-asthmatic Controls: Age-similar controls will undergo diagnostic bronchoscopy for clinical indications in the absence of known asthma, including recurrent pneumonia, congenital lung anomalies, prolonged cough, suspected laryngeal abnormalities, and suspected aspiration syndromes. Inclusion in the final set to be determined post-procedure based on BAL granulocyte profiles. To be included as a control, participants must have pauci-granular BAL counts (less than 2 percent eosinophils and less than 4 percent PMN), no positive allergen sensitization, and no positive viral or bacterial studies from analysis of BAL fluid.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — A diagnostic bronchoscopy will be conducted for clinical indications in children referred to the University of Virginia Children's Hospital for evaluation of respiratory symptoms

SUMMARY:
The pattern of lower airway inflammation in asthma is heterogeneous, but in many patients, the polymorphonuclear neutrophil (PMN) is the predominant granulocyte infiltrating the airspaces. Although it is known to have an important function in innate immune defense, the role of the PMN in asthma has not been well elucidated. In work in progress, the investigators have identified the receptor for IL-5 on the surface of bronchoalveolar lavage (BAL) PMNs in a subset of children with severe, treatment-resistant asthma, a characteristic that is not found in peripheral blood neutrophils. While the function of this IL-5 receptor has yet to be determined, preliminary evidence strongly supports a mechanism linking neutrophilic with type 2 inflammation in the lower airways of children with asthma, a discovery that has exciting potential to modify the treatment of asthma.

The primary objective of this observational cross-sectional study is to test the overall hypothesis that therapeutic intervention directed against the IL-5R on lung PMNs will decrease inflammation and improve clinical outcomes in patients with poorly controlled asthma. The secondary study objective is to demonstrate that IL-5R expression on lung-infiltrating PMNs is functional, will activate known IL-5R-induced signaling pathways, and will lead to enhanced PMN pro-inflammatory activity including increased PMN recruitment, prolonged survival, degranulation, and release of reactive oxygen species.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-17
* Treatment-resistant, refractory respiratory symptoms
* Scheduled for a clinical diagnostic bronchoscopy

Exclusion Criteria:

* Known lower respiratory tract infection within 60 days of scheduled bronchoscopy
* Systemic disorders involving the heart, respiratory system, CNS, renal, and endocrine systems

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes children with refractory respiratory symptoms, most who will have poorly-controlled asthma. An age similar comparison group with structural lung anomalies who undergo diagnostic bronchoscopy will serve as controls.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Percent neutrophils bearing surface markers for IL-5 Receptor | 6+ months post bronchoscopy
  The percentage of neutrophils which bear surface markers for the IL5-R in lung fluid and peripheral blood will be compared in children with different asthma phenotypes

SECONDARY OUTCOMES:
In vitro analysis of IL-5 Receptor (IL-5 R) function: Signaling via the IL-5 R displayed on neutrophils from the BAL (and if necessary, peripheral blood) following ligand (IL-5) binding | 48-72 hours post bronchoscopy
  This measure will assess the phosphorylation of STAT 5 and simultaneously phosphorylation of AKT (as a surrogate for activation of PI 3 kinase) following treatment of neutrophils with IL-5 (i.e. IL-5 R engagement). Engagement of the GM-CSF receptor on the neutrophils by its ligand will serve as a control for the capacity of neutrophils to undergo signal transduction in response to ligands. Additional control will be activation (phosphorylation) of STAT 5 on eosinophils responding to IL-5 (i.e IL-5 R engagement). This analysis will be carried out using flow cytometry to evaluate phosphorylation of the indicated signaling intermediates. This analysis will establish whether the IL-5 R on BAL neutrophils is functional (i.e. capable of transducing a signal following ligand binding).
Measurement of neutrophil degranulation and inflammatory mediator production following IL-5 binding to its receptor on neutrophils isolated from the BAL | 48-72 hours post bronchoscopy
  Neutrophil activation will assess the production of specific cytokines (e.g. TNFa) and chemokines (e.g. CXCL 10) as well as release of granule contents (e.g. lysozyme and proteases) following IL-5 R engagement. These functions will be assessed by ELISA. Analysis of this parameter will elucidate whether signaling through the IL-5 R results in classical activation of IL-5 R positive neutrophils, the result of which is enhanced injury and inflammation.
Production of Reactive Oxygen Species following IL-5 R engagement | 48-72 hours post bronchoscopy
  Reactive Oxygen Species will evaluate the generation of ROS by neutrophils following IL-5 R engagement in BAL neutrophils (and if appropriate neutrophils isolated from peripheral blood). This analysis will be carried out using colorimetric analysis of color change in neutrophils exposed to ROS sensitive dye. This analysis will determine if exposure to IL-5 results in ROS production by neutrophils and as a consequence the potential for increased tissue damage to the lungs.
Measurement of neutrophil survival in culture upon IL-5 R engagement in vitro | 48-72 hours post bronchoscopy
  Neutrophil survival will analyze the survival in culture of neutrophils isolated from the BAL following exposure to IL-5 in vitro. Apoptosis of neutrophils over time in culture will be evaluated by flow cytometry. This analysis will determine whether exposure of lung neutrophils to IL-5 will enhance their survival and therefore the potential of neutrophils activated in response to IL-5 to promote enhanced inflammation and injury.

CONTACTS AND LOCATIONS:
Overall Officials: William G Teague, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No